CLINICAL TRIAL: NCT04568642
Title: Randomized Crossover Trial to Compare Closed-loop FiO2 Controller With Conventional Control of FiO2 During Mechanical Ventilation of Pediatric Patients
Brief Title: Comparing Closed-loop FiO2 Controller With Conventional Control of FiO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Hasan ağın, Professor doctor, Head of pediatric intensive care unit (PICU), Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02020/404
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Failure; Acute Hypoxemic Respiratory Failure; Acute Hypoxemic and Hypercapnic Respiratory Failure
Keywords: Acute respiratory failure (ARF); Pediatric acute respiratory distress syndrome (PARDS),; Acute lung injury (ALI),; SpO2; FiO2
MeSH Terms: conditions — Respiratory Insufficiency; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Device: conventional FiO2 will be selected by the clinician according to the SpO2 target
  Interventions: Device: Deactivate FiO2 controller
- Closed-loop (Experimental): Device: conventional FiO2 will be selected by the closed-loop algorithm according to the SpO2 target
  Interventions: Device: Activate FiO2 controller

INTERVENTIONS:
Device: Activate FiO2 controller — Closed-loop FiO2 controller will be activated in the experimental arm
  Arms: Closed-loop
Device: Deactivate FiO2 controller — Closed-loop FiO2 controller will be deactivated in the experimental arm
  Arms: Conventional

SUMMARY:
During mechanical ventilation (MV) hypoxemic or hyperoxemic events should be carefully monitored and a quick response should be provided by the caregiver at the bedside. Pediatric mechanical ventilation consensus conference (PEMVECC) guidelines suggest to measure SpO2 in all ventilated children and furthermore to measure partial arterial oxygen pressure (PaO2) in moderate-to-severe disease. There were no predefined upper and lower limits for oxygenation in pediatric guidelines, however, Pediatric acute lung injury consensus conference PALICC guidelines proposed SpO2 between 92 - 97% when positive end-expiratory pressure (PEEP) is smaller than 10 cm H2O and SpO2 of 88 - 92% when PEEP is bigger or equal to 10 cm H2O. [1] For healthy lung, PEMVECC proposed the SpO2>95% when breathing a FiO2 of 21%.[2] As a rule of thumb, the minimum fraction of inspired O2 (FiO2) to reach these targets should be used. A recent Meta-analyze showed that automated FiO2 adjustment provides a significant improvement of time in target saturations, reduces periods of hyperoxia, and severe hypoxia in preterm infants on positive pressure respiratory support. [3] This study aims to compare the closed-loop FiO2 controller with conventional control of FiO2 during mechanical ventilation of pediatric patients

DETAILED DESCRIPTION:
The study has a crossover design. Patients will start in standard ASV 1.1 settings, then attending physician will assess the ventilation parameters according to study protocol and will note them in the case report form as he starts the data recording with MemoryBox (MB)in the mixed mode. Afterwards, the clinician will start the first phase by either keeping the patient in ASV 1.1 without any closed-loop controllers activated or switching to ASV 1.1 with only FiO2 controller activated according to the randomization. After 2.5 hours of recording in the first phase, the clinician will switch the patient to the second phase regarding randomization order. If the patient was ventilated without FiO2 controller activated in the first phase, the controller will be activated in the second phase. The patient will stay in the second phase for 2.5 hours as well. The first 0.5 hours of the first phase will be considered as run-in phase and the first 0.5 hours of the second phase will be considered as wash-out phase. Therefore the first 0.5 hours of each phase will be excluded from data analysis due to cross-over study design.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 1 months and 18 years
* Patients above 7kg of IBW
* Informed consent was signed by next of kin
* Requiring FiO2 ≥ 25% to keep SpO2 in the target ranges defined by the clinician

Exclusion Criteria:

* Candidate for extubation in the next 5 hours.
* Patient included in another interventional study in the last 30 days
* Hemodynamically instable patients (defined as a need for continuous infusion of epinephrine or norepinephrine > 1 mg/h)
* Patients with congenital or acquired hemoglobinopathies effecting SpO2 measurement
* Patient included in another interventional research study under consent
* Patient already enrolled in the present study in a previous episode of acute respiratory failure

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
optimum range time | 2 hour
  Percentage of time spent in the defined optimum SpO2 range (percentage)

SECONDARY OUTCOMES:
Acceptable range time | 2 hour
  Percentage of time spent in the defined acceptable SpO2 range (percentage)
Suboptimum range time | 2 hour
  Percentage of time spent in the defined suboptimum SpO2 range (percentage)
Manuel adjustments | 2 hour
  number of FiO2 controller manuel adjustments

CONTACTS AND LOCATIONS:
Locations (1):
- The Health Sciences University Izmir Behçet Uz Child Health and Diseases education and research hospital, Izmir, Turkey/izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santschi M, Jouvet P, Leclerc F, Gauvin F, Newth CJ, Carroll CL, Flori H, Tasker RC, Rimensberger PC, Randolph AG; PALIVE Investigators; Pediatric Acute Lung Injury and Sepsis Investigators Network (PALISI); European Society of Pediatric and Neonatal Intensive Care (ESPNIC). Acute lung injury in children: therapeutic practice and feasibility of international clinical trials. Pediatr Crit Care Med. 2010 Nov;11(6):681-9. doi: 10.1097/PCC.0b013e3181d904c0. PMID 20228688
- [Background] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Background] Kneyber MCJ, de Luca D, Calderini E, Jarreau PH, Javouhey E, Lopez-Herce J, Hammer J, Macrae D, Markhorst DG, Medina A, Pons-Odena M, Racca F, Wolf G, Biban P, Brierley J, Rimensberger PC; section Respiratory Failure of the European Society for Paediatric and Neonatal Intensive Care. Recommendations for mechanical ventilation of critically ill children from the Paediatric Mechanical Ventilation Consensus Conference (PEMVECC). Intensive Care Med. 2017 Dec;43(12):1764-1780. doi: 10.1007/s00134-017-4920-z. Epub 2017 Sep 22. PMID 28936698
- [Background] Mitra S, Singh B, El-Naggar W, McMillan DD. Automated versus manual control of inspired oxygen to target oxygen saturation in preterm infants: a systematic review and meta-analysis. J Perinatol. 2018 Apr;38(4):351-360. doi: 10.1038/s41372-017-0037-z. Epub 2018 Jan 2. PMID 29296004
- [Background] Waitz M, Schmid MB, Fuchs H, Mendler MR, Dreyhaupt J, Hummler HD. Effects of automated adjustment of the inspired oxygen on fluctuations of arterial and regional cerebral tissue oxygenation in preterm infants with frequent desaturations. J Pediatr. 2015 Feb;166(2):240-4.e1. doi: 10.1016/j.jpeds.2014.10.007. Epub 2014 Nov 18. PMID 25454938
- [Background] Dani C. Automated control of inspired oxygen (FiO2 ) in preterm infants: Literature review. Pediatr Pulmonol. 2019 Mar;54(3):358-363. doi: 10.1002/ppul.24238. Epub 2019 Jan 10. PMID 30632296
- [Background] Lal M, Tin W, Sinha S. Automated control of inspired oxygen in ventilated preterm infants: crossover physiological study. Acta Paediatr. 2015 Nov;104(11):1084-9. doi: 10.1111/apa.13137. PMID 26194933
- [Background] Platen PV, Pomprapa A, Lachmann B, Leonhardt S. The dawn of physiological closed-loop ventilation-a review. Crit Care. 2020 Mar 29;24(1):121. doi: 10.1186/s13054-020-2810-1. PMID 32223754
- [Derived] Soydan E, Ceylan G, Topal S, Hepduman P, Atakul G, Colak M, Sandal O, Sari F, Karaarslan U, Novotni D, Schultz MJ, Agin H. Automated closed-loop FiO2 titration increases the percentage of time spent in optimal zones of oxygen saturation in pediatric patients-A randomized crossover clinical trial. Front Med (Lausanne). 2022 Aug 25;9:969218. doi: 10.3389/fmed.2022.969218. eCollection 2022. PMID 36091711